CLINICAL TRIAL: NCT05442710
Title: Recovery From Acute Immune Failure in Septic Shock by Immune Cell Extracorporeal Therapy
Acronym: ReActiF-ICE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Artcline GmbH (Industry)
Collaborators: Zentrum für Klinische Studien Jena (Other); RQM+ (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReActIF-ICE_ZKSJ0124
Record Dates: First submitted 2022-06-07; First posted 2022-07-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled parallel-group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARTICE Treatment Group (Experimental): Subjects with septic shock treated with immune cell extracorporeal therapy on top of standard of care
  Interventions: Biological: ARTICE
- Control Group (No Intervention): Subjects with septic shock receiving standard of care

INTERVENTIONS:
Biological: ARTICE — Extracorporal treatment with purified granulocyte concentrate
  Arms: ARTICE Treatment Group

SUMMARY:
Evaluation of a novel therapy approach for severe sepsis patients. Subjects randomized into the treatment arm receive treatment with an immune cell perfusion system on top of standard care.

This may contribute to the improvement of the impaired organ function of septic shock patients by assisting the impaired immune system (immune competence enhancement = ARTICE)

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects

   1. ≥ 18 years of age
   2. with septic shock, defined as those with septic shock according to" Sepsis-3-Definition" who additionally require norepinephrine at a dose of ≥ 0.15 mcg/kg/min (and/or vasopressin at any dose) for a minimum of 6 hours (within the last 48 hours), to maintain a MAP ≥65 mmHg
   3. Subjects ≥ 80 years of age shall have a Clinical Frailty Scale of <5 to be enrolled.
2. Fulfillment of the definition of septic shock, not longer than 48h before randomization. I.e. the 48h start at the end of the 6h period.
3. Blood lactate >2 mmol/L despite adequate volume resuscitation during the current sepsis episode
4. Source control achieved / in progress in the judgement of the investigator
5. Subjects are required to have central venous access and an arterial line, and these are expected to remain present for at least the initial 48 hours of study.
6. Subjects must have received adequate volume replacement in the judgement of the investigator.
7. Subject or legal surrogate is willing and able to provide written informed consent and comply with all protocol requirements or confirmation of the urgency of participation in the clinical trial and the possible benefit to the subject by an independent consultant or the implementation of other established procedures according to the local regulations of the contributing centre to include subjects who are unable to provide informed consent.

Exclusion Criteria:

1. Acute or chronic leukemia,
2. Bilirubin ≥ 2 mg/dL (≥33 µmol/L),
3. Ongoing (concomitant) or prior within the last 6 month any chemotherapy or radiotherapy for malignancy,
4. Autoimmune disease with systemic medication of ≥10 mg prednisolone equivalent,
5. Previous transplantation,
6. Subjects receiving interferon therapy (14 days prior randomisation),
7. Acute pulmonary embolism within the last 72 hours,
8. Ischemic stroke or intracranial bleeding within the last 3 months
9. Suspicion of concomitant acute coronary syndrome based on clinical symptoms and/or ECG within the last 72 hours,
10. Cardiopulmonary resuscitation within last 7 days,
11. Moribund subject (life expectancy <72 hours), in the judgement of the investigator
12. Presence of a do-not-resuscitate or do-not-intubate order,
13. Known HIV infection or chronic viral hepatitis,
14. Isolated Urosepsis,
15. Pregnancy/nursing period,
16. Primary cause of hypotension not due to sepsis (e.g. major trauma including traumatic brain injury, haemorrhage, burns, or congestive heart failure/cardiogenic shock),
17. Previous sepsis with ICU admission within this hospital stay,
18. Known/suspected acute mesenteric ischaemia,
19. Chronic mechanical ventilation for any reason OR severe COPD requiring either continuous daily oxygen use during the preceding 30 days or mechanical ventilation (for acute exacerbation of COPD) during the preceding 30 days,
20. Decision to limit full care taken before obtaining informed consent,
21. Prior enrolment in the trial,
22. Prior use of an investigational medicinal product within the last month OR planned or concurrent participation in a clinical trial for any investigational drug or device,
23. multiple injuries including polytrauma and burn >20% TBSA (2° or 3°),
24. Diagnosed and documented pre-existing dementia,
25. Severe Covid-Pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-07-24 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the ARTICE therapy, composed of new onset of serious adverse events from re-evaluation on Day 2 through Day 28 | From re-evaluation on Day 2 through Day 28
  The number [n] of new onsets of serious adverse events (SAEs) from re-evaluation-Day 2 through Day 28 will be counted in both arms and the difference between groups will be compared.

SECONDARY OUTCOMES:
All cause mortality through Day 28 | From re-evaluation on Day 2 through Day 28
  The difference in all-cause mortality from re-evaluation on Day 2 through Day 28 will be measured by time to event and Relative risk as well as Kaplan-Meier estimates with 95%-CI will be calculated through day 28
All cause mortality through Day 90 | From re-evaluation on Day 2 through Day 90
  The difference in all-cause mortality from re-evaluation on Day 2 through Day 90 will be measured by time to event and Relative risk as well as Kaplan-Meier estimates with 95%-CI will be calculated through day 90
All-cause in-hospital mortality | From re-evaluation on Day 2 through until hospital discharge
  The difference in all-cause mortality from re-evaluation on Day 2 through hospital discharge will be measured by time to event and Relative risk as well as Kaplan-Meier estimates with 95%-CI will be calculated through hospital discharge.
Daily changes in total SOFA and SOFA sub-scores | Until Day 10
  The SOFA (Sequential organ failure assessment score) Score URL"Sequential Organ Failure Assessment (SOFA) Score - MDCalc" is measured by addition of 6 Subscores for each of the 6 Organs between 1 and 4 [n]. The Change from Baseline (COBL) inbetween groups will be compared daily until day 10.
  Total score ranges from 0 (best) to 24 (worst); Subscores range from 0 (best) to 4 (worst)
Time course of key inflammatory/ immunological markers in between the two groups. | From re-evaluation on Day 2 until Day 28
  Time course of key inflammatory/ immunological markers including mHLA-DR and cytokines, measured by their concentration in plasma in pg/mL or in % (HLA-DR) until day 28. Their plasma concentration will be compared by each day inbetween groups.
Time to complete organ failure resolution | From re-evaluation on Day 2 until Day 28 with special focus on D14 an D21
  The Time to complete organ failure resolution of the 6 organs of the SOFA system (measured as the time from a Baseline value>1 until the score/subscore is 0) through Day 14 and Day 21 will be measured and the time to resolution for all failed organs as a Kaplan Meier Model.
ICU length of stay Measured / Confirmed on day 28 retrospectively. Units: Days | Until Day 28
  ICU length of stay (through Day 28) will be measured as days [n] in the ICU and compared in between the groups
Number of hospital-free days. Measured / Confirmed on day 28 retrospectively. Units: Days | Until Day 28
  Hospital length of stay and number of hospital-free days (through Day 28), measured by number of days [n] will be compared between groups Units: Days
Number of ICU-free days Measured / Confirmed on day 28 retrospectively. Units: Days | Until day 28
  ICU length of stay and number of ICU-free days (through Day 28), measured by number of days [n] will be compared between groups Units: Days
Number of vasopressor- free days | From re-evaluation on Day 2 until Day 28
  Number of vasopressor- free days [n], until Day 28 Measured / Confirmed on day 28 retrospectively. Units: Days
Number of mechanical-ventilator-free days | From re-evaluation on Day 2 until Day 28
  Number of mechanical-ventilator-free days [n], until Day 28 Measured / Confirmed on day 28 retrospectively. Units: Days
Number of renal-replacement-free days | From re-evaluation on Day 2 until Day 28
  Number of renal-replacement-free days [n] until Day 28. Measured / Confirmed on day 28 retrospectively. Units: Days
Number of days without antimicrobial therapy | From re-evaluation on Day 2 until Day 28
  Number of days [n] without antimicrobial therapy, until Day 28. Measured / Confirmed on day 28 retrospectively. Units: Days
Frequency of secondary infections | From re-evaluation on Day 2 until Day 28
  Frequency of secondary infections [n], until Day 28. Measured / Confirmed on day 28 retrospectively. Units: total number and days
Antibiotic exposure days until hospital discharge | From re-evaluation on Day 2 until Day 28
  Antibiotic exposure days [n] until hospital discharge (maximum until Day 28). Measured / Confirmed on day 28 retrospectively. Units: Days
Days [n] alive without antibiotics until hospital discharge | From re-evaluation on Day 2 until Day 28
  Days alive without antibiotics until hospital discharge (maximum until Day 28). Measured / Confirmed on day 28 retrospectively. Units: Days
Total daily dose of noradrenalin (NA) administered on each day | From re-evaluation on Day 2 until Day 10
  Total daily dose of noradrenalin (NA) administered on each day measured in mg/kg between Day 2 and Day 10 will be compared in between groups.
Maximum daily dose of noradrenalin administration on treatment days | From re-evaluation on Day 2 until Day 10
  Maximum daily dose of noradrenalin administration on treatment days between Day 2 and Day 10 (applied for a minimum of 30 min) will be measured as µg/kg/min and compared between the groups for each day until day 10.
Occurrence of virus induced inflammation episodes | From re-evaluation on Day 2 until Day 28
  Occurrence of virus induced inflammation episodes, especially reactivation of CMV, HSV etc. will be counted as an (S)AE until 28 and the number [n] will be compared between groups.
  Measured / Confirmed on day 28 retrospectively.
Quality of life assessment | Until day 90
  Quality of life assessed at baseline, Day 28 and Day 90 using EQ-5D-5L Score [n] and compared between the groups.
  EQ-5D-5L' is not an abbreviation, it can be described as "EuroQuol - 5 Dimensions - 5 Levels". It considers five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression at 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers result in a 1-digit number for each dimension. The digits (1= no problem to 5=extreme problems) can be combined into a 5-digit number that describes the patient's health state. 11111 indicates no problems on any of the five dimensions.
  The EQ VAS visual analogue scale records the patient's self-rated health. The endpoints are labelled 'The best health you can imagine' (=100) and 'The worst health you can imagine' (=0).
Occurrence of cognitive decline | Until day 90
  Occurrence of cognitive decline at Day 90 compared with baseline and between groups (measured by IQCODE (Questionnaire on cognitive decline in the elderly); [n]) will be compared between groups.
  The IQCODE is scored by averaging the ratings across 26 everyday situations. A person without cognitive decline will have an average score of 3, while scores above 3 indicate that some decline has occurred
Time course of key biomarkers of neuroaxonal injury | Until day 28
  Time course of key biomarkers of neuroaxonal injury (pg/ml) will be measured in the blood of study patients at predefined time points to assess changes in biomarker levels longitudinally over the course of the disease by comparing them in between groups daily.
Inflammatory mRNA profiling analysis | until day 10
  In patients, giving extra informed consent, inflammatory mRNA profiling measured by mRNA occurrence will be analyzed at Day 2 and Day 10 and compared in between Groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Reuter, Prof.Dr., Principal Investigator — University Hospital Rostock
Locations (20):
- Germany (20):
  - Universitätsklinikum Freiburg, Interdisziplinäre Medizinische Intensivtherapie (IMIT), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Klinik für Anästhesiologie, Regensburg, Bavaria
  - Universitätsklinikum Bonn, Klinik und Poliklinik für Anästhesiologie und Operative Intensivmedizin, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Köln, Klinik für Anästhesiologie und Operative Intensivmedizin, Cologne, North Rhine-Westphalia
  - Helios Klinikum Aue, Aue, Saxony
  - Universitätsklinikum Leipzig, Klinik und PK für Anästhesiologie und Intensivtherapie, Leipzig, Saxony
  - Universitätsklinikum Halle (Saale), Universitätsklinik für Anästhesiologie und Operative Intensivmedizin, Halle, Saxony-Anhalt
  - UNIVERSITÄTSKLINIKUM Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Charité Berlin, Klinik mit Schwerpunkt Nephrologie und internistische Intensivmedizin, Berlin
  - Klinikum Braunschweig, Medizinische Klinik V, Braunschweig
  - Universitätsklinikum Essen, Klinik für Nephrologie, Essen
  - University Hospital Frankfurt, Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, Frankfurt
  - Helios Klinikum HIldesheim, Hildesheim
  - Klinikum Magdeburg, Klinik für Intensiv- und Rettungsmedizin, Magdeburg
  - University Medical Center Mainz, Study center for Anesthesiology, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - University Hospital Minden, Departmenr of Anaesthesiology, intensive and emergency care, Minden
  - Klinikum Oldenburg, Universitätsklinik für Anästhesiologie/ Intensivmedizin, Oldenburg
  - Universitätsmedizin Rostock, Abteilung KAI, Rostock
  - Helios Kliniken Schwerin, Department for intensive care, Schwerin

IPD SHARING:
Plan to Share IPD: No